CLINICAL TRIAL: NCT05726864
Title: First in Human Phase 1/2 Trial of ELI-002 7P Immunotherapy as Treatment for Subjects With Kirsten Rat Sarcoma (KRAS)/Neuroblastoma RAS Viral Oncogene Homolog (NRAS) Mutated Pancreatic Ductal Adenocarcinoma (PDAC) and Other Solid Tumors
Brief Title: A Study of ELI-002 7P in Subjects With KRAS/NRAS Mutated Solid Tumors
Acronym: AMPLIFY-7P
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Elicio Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ELI-002-201
Record Dates: First submitted 2023-02-03; First posted 2023-02-14 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Pancreatic Ductal Adenocarcinoma; Colorectal Cancer; KRAS G12D; KRAS G12R; KRAS G12V; KRAS G12A; KRAS G12C; KRAS G12S; KRAS G13D; NRAS G12D; NRAS G12R; NRAS G12V; NRAS G12C; NRAS G12S
Keywords: Kirsten rat sarcoma (KRAS); Neuroblastoma ras viral oncogene homolog (NRAS); Pancreatic ductal adenocarcinoma (PDAC); Colorectal cancer (CRC); Colon cancer; Rectal cancer; Immunotherapy; Vaccine therapy; Adjuvant therapy; serum tumor biomarker; Carbohydrate antigen 19-9 (CA19-9); Carcinoembryonic antigen (CEA); circulating tumor DNA (ctDNA)
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase 1A: ELI-002 7P (Low Peptide dose) (Experimental): ELI-002 Amph-CpG-7909 (10.0mg) admixed with ELI-002 Amph-Peptides 7P (1.4mg) administered via SC injection weekly for 4 consecutive weeks, followed by bi-weekly injections over 4 weeks, during the Immunization Period; additional SC injections for 4 consecutive weeks during the Booster Period (the two periods are separated by 2 months of no dosing)
  Interventions: Drug: ELI-002 7P
- Phase 1A: ELI-002 7P (High Peptide dose) (Experimental): ELI-002 Amph-CpG-7909 (10.0mg) admixed with ELI-002 Amph-Peptides 7P (4.9mg) administered via SC injection weekly for 4 consecutive weeks, followed by bi-weekly injections over 4 weeks, during the Immunization Period; additional SC injections for 4 consecutive weeks during the Booster Period (the two periods are separated by 2 months of no dosing)
  Interventions: Drug: ELI-002 7P
- Phase 1B: ELI-002 7P (Experimental): The ELI-002 7P dose selected during the Phase 1A portion of the study will be administered via SC injection weekly for 4 consecutive weeks, followed by bi-weekly injections over 4 weeks, during the Immunization Period; additional SC injections for 4 consecutive weeks during the Booster Period (the two periods are separated by 2 months of no dosing)
  Interventions: Drug: ELI-002 7P
- Phase 2 randomized: ELI-002 7P (Experimental): The ELI-002 7P dose selected during the Phase 1A portion of the study will be administered via SC injection weekly for 4 consecutive weeks, followed by bi-weekly injections over 4 weeks, during the Immunization Period; additional SC injections for 4 consecutive weeks during the Booster Period (the two periods are separated by 2 months of no dosing)
  Interventions: Drug: ELI-002 7P

INTERVENTIONS:
Drug: ELI-002 7P — ELI-002 Amph-CpG-7909 admixed with ELI-002 Amph-Peptides 7P administered via SC injection weekly for 4 consecutive weeks, followed by bi-weekly injections over 4 weeks, during the Immunization Period; additional SC injections weekly for 4 weeks during the Booster Period (the two periods are separated by 2 months of no dosing)

SUMMARY:
This is a Phase 1/2 study to assess the safety and efficacy of ELI-002 7P immunotherapy (a lipid-conjugated immune-stimulatory oligonucleotide [Amph-CpG-7909] plus a mixture of lipid-conjugated peptide-based antigens [Amph-Peptides 7P]) as adjuvant treatment in subjects with solid tumors with mutated KRAS/NRAS. This study builds on the experience obtained with related product ELI-002 2P, which was studied in protocol ELI-002-001 under IND 26909.

DETAILED DESCRIPTION:
The study consists of 3 phases: Phase 1A, Phase 1B, and Phase 2. In Phase 1A, seven Amph modified KRAS and NRAS peptides, G12D, G12R, G12V, G12A, G12C, G12S, G13D (Amph-Peptides 7P) will be evaluated in combination with recommended Phase 2 dose of Amph-CpG-7909 (10.0mg). This Amph-CpG-7909 dose will be evaluated with two Amph-Peptides 7P dose levels (1.4mg and 4.9mg) in 6 subjects per dose level. Following enrollment of these 12 subjects, the independent data monitoring committee (IDMC) will decide if another 6 subjects should be enrolled or if the dose can be determined for Phase 1B and Phase 2 portions of the study to be opened. If another 6 subjects are enrolled to Phase 1A, the IDMC will meet again to decide upon the dose for Phase 1B and Phase 2 prior to opening these portions of the study.

In Phase 1B, one dose expansion cohort of up to 17 colorectal cancer [CRC] subjects may be added to evaluate for preliminary evidence of biomarker response, including circulating tumor deoxyribonucleic acid (ctDNA) and/or serum tumor biomarker (such as CA19-9 and CEA) reduction and clearance in KRAS and NRAS.

In Phase 2, an additional 135 PDAC subjects will be randomized 2:1 (ELI-002 7P versus observation) to further evaluate antitumor activity. Subjects randomized to ELI-002 7P will receive subcutaneous (SC) injections of ELI-002 7P during Immunization and Booster Periods. Subjects randomized to observation will have the same safety and efficacy evaluations and will follow the same assessment schedule as subjects randomized to ELI-002 7P but will not receive study treatment. Subjects randomized to observation will be able to elect to cross-over to ELI-002 7P treatment in the event of confirmed disease progression.

ELIGIBILITY:
Inclusion Criteria:

* KRAS/NRAS mutated (G12D, G12R, G12V, G12A, G12C, G12S, G13D) solid tumor
* Phase 1 only: positive for circulating tumor DNA and/or elevated serum tumor biomarkers (such as CA19-9 and CEA) despite prior standard therapy including surgery and chemotherapy/radiation therapy where applicable
* Screening CT is negative for recurrent disease
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1

Exclusion Criteria:

* Presence of tumor mutations where specific therapy is approved
* Known brain metastases
* Use of immunosuppressive drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2023-04-14 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Evaluate the safety of ELI-002 7P | 28 days after the first dose of ELI-002 7P
  Safety will be assessed by the incidence of adverse events (AEs) and clinically significant changes in laboratory tests and vital signs
Phase 2: Compare ELI-002 7P versus standard of care (SOC; observation) in DFS (disease free survival) | After the last radiographic assessment at Visit 26 (Week 150)
  DFS is assessed by the investigator through computed tomography (CT) imaging or magnetic resonance imaging (MRI) with contrast and using iRECIST criteria

SECONDARY OUTCOMES:
Phase 2: Overall Survival (OS) | After Visit 13 (Week 20)
  To compare OS between cohorts, ELI-002 7P vs Observation
Phase 1 and Phase 2: Determine the biomarker reduction or clearance rate | 6 months
  The ctDNA reduction or clearance is defined as reduction or clearance of ctDNA from baseline, or if ctDNA was not detectable at baseline, serum tumor biomarker (such as CA19-9 and CEA) reduction and clearance compared to baseline
Phase 2: Determine the 1-year DFS | 1 year
  Compare between cohorts, ELI-002 7P vs Observation, the 1-year DFS
Phase 2: Evaluate the safety of ELI-002 7P | 30 days after the last ELI-002 7P dose
  Safety will be assessed by the incidence of AEs and clinically significant laboratory tests and vital signs

CONTACTS AND LOCATIONS:
Locations (28):
- United States (28):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Mayo Clinic Comprehensive Cancer Center, Phoenix, Arizona
  - City of Hope, Duarte, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California Los Angeles, Los Angeles, California
  - University of California, Irvine, Orange, California
  - University of Colorado Hospital-Anschutz Cancer Pavillion, Aurora, Colorado
  - University of Miami, Coral Gables, Florida
  - University of Florida Health Cancer Center, Gainesville, Florida
  - Mayo Clinic Comprehensive Cancer Center, Jacksonville, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Emory Winship Cancer Institute, Atlanta, Georgia
  - University of Iowa, Iowa City, Iowa
  - Ochsner Health, New Orleans, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic Comprehensive Cancer Center, Rochester, Minnesota
  - Northwell Health, Lake Success, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - New York Presbyterian Weill Cornell Medical Center, New York, New York
  - Lehigh Valley Health Network, Allentown, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Southwestern, Dallas, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin